CLINICAL TRIAL: NCT07233161
Title: Effectiveness of m-CIMT of the Upper Limb in Acute Post-stroke Patients.
Brief Title: Effectiveness of m-CIMT of the Upper Limb in Acute Post-stroke Patients. (m-CIMT, Modified Constraint-induced Movement Therapy)
Acronym: m-CIMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2024/1353
Record Dates: First submitted 2025-06-05; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Isquemic Stroke; Upper Limb Weakness Due to Central Neurologic Injury
Keywords: m-CIMT; stroke; upper limb weakness; upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomised, single-centre, single-blind, prospective, prospective clinical trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): m-CIMT therapy
  Interventions: Behavioral: m-CIMT
- Control group (No Intervention): Conventional treatment

INTERVENTIONS:
Behavioral: m-CIMT — m-CIMT therapy (healthy side restraint) and a specific upper limb exercise protocol.
  Other Names: m-CIMT protocol
  Arms: Experimental

SUMMARY:
m-CIMT therapy is the restriction of the unaffected upper extremity in conjunction with an upper extremity specific exercise protocol to improve the functionality and use of the affected upper extremity.

DETAILED DESCRIPTION:
The study consists of a total of 7 days with a total of 3 hours per day of restraint of the unaffected upper limb together with 1 physiotherapy session per day specific to the affected upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic stroke.
* Hospitalised patient (first 15 days).
* Ability to understand and execute simple instructions.
* Over 18 years of age.
* Upper limb motor deficit.
* Sign the informed consent document.

Exclusion Criteria:

* Unstable clinical/medical condition.
* Limitation of the upper limb due to a previous stroke.
* Strokes affecting both upper limbs bilaterally.
* Fractures/dislocations in the joints of the affected upper limb that may affect recovery.
* Severe behavioural disturbance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer | Basal, immediately after the intervention, 3 months after treatment
  The Fugl-Meyer Upper Extremity Scale assesses motor function of the arm and hand after stroke. It measures movements, reflexes and coordination, with a maximum score of 66. It is a structure-measuring tool. This scale is scored from 0 to 66 with 66 being the best score.
Abilhand | Basal, immediately after the intervention, 3 months after treatment
  The ABILHAND assesses a person's ability to perform manual activities of daily living. It is based on the patient's perception of the difficulty of these tasks. It is a tool for measuring activity. This scale is scored from 0 to 46 with 46 being the best score.
Motor Activity Log | 3 months after treatment
  The Motor Activity Log (MAL) assesses how much and how well a person uses their affected arm in everyday activities after a stroke. It is based on interviews and rates the Amount of Use and Quality of Movement of the use of the paretic arm in daily life. This scale has two scores, quality and quantity. From 0 to 150 for quantity and from 0 to 150 for quality. 150 being the best result in both cases.
Fatigue Assessment Scale (FAS) | Basal, immediately after the intervention, 3 months after treatment
  The Fatigue Assessment Scale (FAS) is a questionnaire that assesses the level of physical and mental fatigue in patients with various health conditions. It consists of 10 items that the patient answers according to their recent experience.
  This scale has two scores: Mental fatigue from 0 to 25 (sum of items 3, 6, 7, 8 and 9) and physical fatigue from 0 to 25 (sum of items 1, 2, 4, 5 and 10). With 25 being the worst score for both cases.
Stroke Impact Scale | Basal,immediately after the intervention, 3 months after treatment
  The Stroke Impact Scale (SIS) assesses the difficulty a person has in performing daily activities during the last two weeks after a stroke. The minimum score on this scale is 16 points and the maximum is 80 points, with 80 being the best score.

SECONDARY OUTCOMES:
Modified Rankin Scale (MRS) | Basal, immediately after the intervention, 3 months after treatment
  The modified Rankin Scale (MRS) assesses the degree of disability or dependence in daily activities after a stroke. It ranges from 0 (no symptoms) to 6 (death). The minimum score is 0 and the maximum score is 5 points. The worst score is 5 points.
National Institutes of Health Stroke Scale (NIHSS) | Basal, immediately after the intervention, 3 months after treatment
  The NIHSS (National Institutes of Health Stroke Scale) is a clinical scale that assesses the severity of stroke. It measures functions such as level of consciousness, language, vision, vision, strength, sensation and coordination. This scale is scored from 0 to 42 with 42 being the worst score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We don't have the url with the information

REFERENCES:
- [Background] Kwakkel G, Veerbeek JM, van Wegen EE, Wolf SL. Constraint-induced movement therapy after stroke. Lancet Neurol. 2015 Feb;14(2):224-34. doi: 10.1016/S1474-4422(14)70160-7. PMID 25772900
- [Background] Thrane G, Askim T, Stock R, Indredavik B, Gjone R, Erichsen A, Anke A. Efficacy of Constraint-Induced Movement Therapy in Early Stroke Rehabilitation: A Randomized Controlled Multisite Trial. Neurorehabil Neural Repair. 2015 Jul;29(6):517-25. doi: 10.1177/1545968314558599. Epub 2014 Nov 14. PMID 25398726
- [Background] Yadav RK, Sharma R, Borah D, Kothari SY. Efficacy of Modified Constraint Induced Movement Therapy in the Treatment of Hemiparetic Upper Limb in Stroke Patients: A Randomized Controlled Trial. J Clin Diagn Res. 2016 Nov;10(11):YC01-YC05. doi: 10.7860/JCDR/2016/23468.8899. Epub 2016 Nov 1. PMID 28050492
- [Background] Corbetta D, Sirtori V, Castellini G, Moja L, Gatti R. Constraint-induced movement therapy for upper extremities in people with stroke. Cochrane Database Syst Rev. 2015 Oct 8;2015(10):CD004433. doi: 10.1002/14651858.CD004433.pub3. PMID 26446577
- [Background] Singh P, Pradhan B. Study to assess the effectiveness of modified constraint-induced movement therapy in stroke subjects: A randomized controlled trial. Ann Indian Acad Neurol. 2013 Apr;16(2):180-4. doi: 10.4103/0972-2327.112461. PMID 23956560